CLINICAL TRIAL: NCT01068678
Title: A Trial Comparing Efficacy and Safety of NN1250 and Insulin Glargine in Subjects With Type 2 Diabetes (BEGIN™: EASY AM)
Brief Title: Comparison of NN1250 With Insulin Glargine in Subjects With Type 2 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3724; 2009-011398-33 (EudraCT Number); U1111-1113-2412 (Other: WHO)
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2015-12-28 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg 3 times weekly (3TW) (Experimental)
  Interventions: Drug: insulin degludec
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously (under the skin) three times weekly. Dose was individually adjusted.
  Arms: IDeg 3 times weekly (3TW)
Drug: insulin glargine — Injected subcutaneously (under the skin) once daily. Dose was individually adjusted.
  Arms: IGlar OD

SUMMARY:
This trial is conducted in Africa, Asia, Europe, and North America. The aim of this clinical trial is to compare the efficacy and safety of NN1250 (insulin degludec (IDeg)) with insulin glargine (IGlar) in subjects with type 2 diabetes currently treated with metformin alone or with metformin combined with an oral anti-diabetic drug (OAD) qualifying for intensified treatment.

ELIGIBILITY:
Inclusion Criteria:

* Insulin naïve subject (allowed are: previous short term insulin treatment up to 14 days; Treatment during hospitalisation or during gestational diabetes is allowed for periods longer than 14 days)
* Current treatment: metformin monotherapy or metformin in any combination with insulin secretagogues (sulphonylurea (SU) or glinide), DPP-4 inhibitor, alpha-glucosidase-inhibitor (acarbose) with unchanged dosing for at least three months prior to Visit 1 with the minimum doses stated: -Metformin: alone or in combination (including fixed combination) 1500 mg daily or maximum tolerated dose (at least 1000 mg daily) -Insulin secretaguogue (sulfonylurea or glinide): minimum half of the daily maximal dose according to local labelling -DPP-4 inhibitor: minimum half of the daily maximal dose according to local labelling -alpha-glucosidase-inhibitor (acarbose): minimum half of the daily maximal dose or maximum tolerated dose
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis
* Body Mass Index (BMI) below or equal to 45.0 kg/m^2

Exclusion Criteria:

* Use within the last 3 months prior to Visit 1 of: thiazoledinediones, exenatide or liraglutide
* Cardiovascular disease, within the last 6 months prior to Visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements (for UK: adequate contraceptive measures are defined as established use of oral, injected or implanted hormonal methods of contraception, sterilisation, intrauterine device or intrauterine system, or consistent use of barrier methods)
* Cancer and medical history of cancer hereof (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (96):
- United States (56):
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Paramount, California
  - Novo Nordisk Investigational Site, Santa Ana, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Perry, Georgia
  - Novo Nordisk Investigational Site, Olympia Fields, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Fishers, Indiana
  - Novo Nordisk Investigational Site, Franklin, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Interlochen, Michigan
  - Novo Nordisk Investigational Site, Jackson, Mississippi
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Lincoln, Nebraska
  - Novo Nordisk Investigational Site, Hamilton, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Canton, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Pottstown, Pennsylvania
  - Novo Nordisk Investigational Site, Upper St.Clair, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Fredericksburg, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Menomonee Falls, Wisconsin
- Canada (13):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Greater Sudbury, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Mirabel, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
  - Novo Nordisk Investigational Site, St. John's
- Czechia (5):
  - Novo Nordisk Investigational Site, Brandýs nad Labem
  - Novo Nordisk Investigational Site, Mladá Boleslav
  - Novo Nordisk Investigational Site, Ostrava
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Trutnov
- Israel (5):
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rehovot
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
  - Novo Nordisk Investigational Site, Safed
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Novo Nordisk Investigational Site, Manatí, Puerto Rico
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Moldava nad Bodvou
  - Novo Nordisk Investigational Site, Nové Zámky
  - Novo Nordisk Investigational Site, Prešov
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
- United Kingdom (9):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Aldershot
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Chippenham
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Nuneaton
  - Novo Nordisk Investigational Site, Portsmouth
  - Novo Nordisk Investigational Site, Watford

REFERENCES:
- [Result] Zinman B, DeVries JH, Bode B, Russell-Jones D, Leiter LA, Moses A, Johansen T, Ratner R; NN1250-3724 (BEGIN:EASY AM) and NN1250-3718 (BEGIN:EASY PM) Trial Investigators. Efficacy and safety of insulin degludec three times a week versus insulin glargine once a day in insulin-naive patients with type 2 diabetes: results of two phase 3, 26 week, randomised, open-label, treat-to-target, non-inferiority trials. Lancet Diabetes Endocrinol. 2013 Oct;1(2):123-31. doi: 10.1016/S2213-8587(13)70013-5. Epub 2013 Jul 9. PMID 24622318
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 94 sites in 7 countries: Canada (14 sites), Czech Republic (5 sites), Israel (5 sites), Slovakia (5 sites), South Africa (3 sites), United Kingdom (8 sites) and United States (54 sites). In addition, 9 sites (United Kingdom (1 site) and United States (8 sites)) were approved, but did not enroll any subjects.
Groups:
- IDeg 3TW: Insulin degludec (IDeg) 200U/mL given 3 times weekly (Mondays, Wednesdays, Fridays) in the morning with metformin with or without dipeptidyl peptidase-4 (DPP-4) inhibitor treatment for 26 weeks.
- IGlar OD: Insulin glargine (IGlar) 100U/mL given once a day (OD), according to the labelling instructions with metformin with or without dipeptidyl peptidase-4 (DPP-4) inhibitor treatment for 26 weeks.
Period: Overall Study
Arm/Group | IDeg 3TW | IGlar OD
Started | 230 | 230
Exposed | 227 (Three subjects withdrew prior to exposure to trial product.) | 229 (one subject withdrew prior to exposure to trial product)
Completed | 192 | 206
Not Completed | 38 | 24
Not completed — Lack of Efficacy | 3 | 2
Not completed — Protocol Violation | 5 | 1
Not completed — Withdrawal criteria | 12 | 6
Not completed — Unclassified | 18 | 15

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)- included all randomised subjects. 1 subject was randomised despite being a screening failure
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg 3TW | IGlar OD | Total
Number analyzed (Participants) | 229 | 230 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.9) | 57.9 (9.7) | 58.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 93 | 198
  Male | 124 | 137 | 261
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.2 (0.8) | 8.3 (0.9) | 8.2 (0.8)
Body weight [Mean (Standard Deviation); unit: kg] | 90.8 (18.6) | 95.7 (19.0) | 93.3 (18.9)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mmol/L] | 9.3 (2.4) | 9.6 (2.4) | 9.5 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after week 26
Time Frame: Week 26
Population: The Full analysis set (FAS) included all randomised subjects and missing data is imputed using last observation carried forward (LOCF).1 subject was randomised despite being a screening failure.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg 3TW | IGlar OD
Number analyzed (Participants) | 229 | 230
percentage of glycosylated haemoglobin | -1.00 (0.95) | -1.40 (1.07)

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline in body weight after week 26
Time Frame: Week 26
Population: The Safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator. Missing data is imputed using last observation carried forward (LOCF). For 3 subjects baseline values were missing.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDeg 3TW | IGlar OD
Number analyzed (Participants) | 227 | 229
kg | 0.8 (3.6) | 1.0 (3.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a time frame of 26 weeks + 7 days follow up
Description: The safety analysis set includes all subjects who received atleast one dose of investigational product or its comparator. 227 subjects in IDeg 3TW and 229 in IGLar OD were included in the analysis.
Arm/Group | IDeg 3TW | IGlar OD
Serious Adverse Events (participants affected / at risk) | 11/227 | 4/229
Other Adverse Events (participants affected / at risk) | 69/227 | 77/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg 3TW (N=227) | IGlar OD (N=229)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg 3TW (N=227) | IGlar OD (N=229)
Diarrhoea (Gastrointestinal disorders) | 16 (17) | 17 (20)
Nausea (Gastrointestinal disorders) | 12 (12) | 15 (16)
Injection site haematoma (General disorders) | 11 (15) | 12 (12)
Nasopharyngitis (Infections and infestations) | 15 (16) | 17 (18)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 16 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (18) | 14 (21)
Headache (Nervous system disorders) | 26 (38) | 21 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.